CLINICAL TRIAL: NCT03659773
Title: A Prospective Cohort Study of Efficacy, Safety and Characterization of Immune Response to Vaccinations in Hematopoietic Stem Cell Transplant Recipients
Brief Title: Immune Response to Vaccinations in Hematopoietic Stem Cell Transplant Recipients
Acronym: VaccHemInf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL17_0769; 2017-A03230-53 (Other: ANSM)
Record Dates: First submitted 2018-07-25; First posted 2018-09-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Vaccination; Hematopoietic Stem Cells
Keywords: Hematopoietic stem cell transplantation; allogeneic hematopoietic stem cell transplantation; autologous hematopoietic stem cell transplantation; vaccination; vaccines; immune function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hematopoietic stem cell transplant (HSCT) (Experimental): immune biomarkers to evaluate vaccine response in HSCT recipients
  Interventions: Biological: immune biomarkers to evaluate vaccine response in HSCT recipients

INTERVENTIONS:
Biological: immune biomarkers to evaluate vaccine response in HSCT recipients — a 38mL-blood sample will be collected before and at 3, 12 and 24 months after complete block vaccination and at 4 weeks after influenza vaccination for the ancillary study

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) is a cellular therapy aiming at curing some hematological diseases. Upon transplantation, recipients experience a phase of profound immune suppression with loss of protective immunity against most infectious agents. Revaccination of HSCT recipients against vaccine-preventable infections is an important post-transplant intervention for reducing morbi-mortality. The VaccHemInf project aims at assessing the efficacy of recommended vaccines in adult recipients of HSCT, through the antibody titers reference method and a panel of immune functional assays.

ELIGIBILITY:
Inclusion Criteria:

* allogeneic and autologous HSCT recipients
* ≥ 18 year-old
* patients having been informed of the conditions of the study (24-month follow-up) and having signed the informed consent form
* Person with social security insurance

  • Additional inclusion criteria for healthy volunteers enrolled (10 volunteers)in the ancillary study of influenza vaccine response:
* health-care workers recruited from the hospital staff

Exclusion Criteria:

* Patient with innate or acquired immune deficiency (severe combined immunodeficiency, Hepatitis C virus (HCV), HBV, HIV infections at any stage)
* Pregnant or breastfeeding women
* History of previous severe allergic reaction to vaccine components
* Patient with no social security coverage, with restricted liberty or under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
proportion of responders defined by the increase in specific antibody titers at 3 months after full block vaccination including tetanus, diphtheria, Pneumococcus, Haemophilus influenza type B (Hib), and hepatitis B virus (HBV). | at 3 months after block vaccination
  ELISA methods will be used to measure serum level concentrations of specific immunoglobulin G (IgG) antibodies to tetanus toxoid, diphtheria toxoid, Hib, pneumococcal capsular polysaccharides and HBV. For pneumococcus, a 4-fold increase in the IgG titer will be considered significant for immunization. For Hib, the values between 0.15-1 μg/mL will be significant for immunization (linearity limit of 9 μg/mL). An IgG titer equal or higher than 0.1 IU/mL for diphtheria and tetanus and higher than 10 mIU/mL for HBV (anti-HBs antibody titer will be considered protective) . An anti-HBs titer higher than 100 IU/mL will be considered to confer long-lasting protection.

SECONDARY OUTCOMES:
proportion of responders defined by the increase in specific antibody titers at 12 months after full block vaccination including tetanus, diphtheria, Pneumococcus, Haemophilus influenza type B (Hib), and hepatitis B virus (HBV). | at 12 months after block vaccination
  ELISA methods will be used to measure serum level concentrations of specific IgG antibodies to tetanus toxoid, diphtheria toxoid, Hib, pneumococcal capsular polysaccharides and HBV. For pneumococcus, a 4-fold increase in the IgG titer will be considered significant for immunization. For the Hib, the values between 0.15-1 μg/mL will be significant for immunization (linearity limit of 9 μg/mL). An IgG titer equal or higher than 0.1 IU/mL for diphtheria and tetanus and higher than 10 mIU/mL for HBV (anti-HBs antibody titer) will be considered protective. An anti-HBs titer higher than 100 IU/mL will be considered to confer long-lasting protection
proportion of responders defined by the increase in specific antibody titers at 24 months after full block vaccination including tetanus, diphtheria, Pneumococcus, Haemophilus influenza type B (Hib), and hepatitis B virus (HBV). | at 24 months after block vaccination
  ELISA methods will be used to measure serum level concentrations of specific IgG antibodies to tetanus toxoid, diphtheria toxoid, Hib, pneumococcal capsular polysaccharides and HBV. For pneumococcus, a 4-fold increase in the IgG titer will be considered significant for immunization. For the Hib, the values between 0.15-1 μg/mL will be significant for immunization (linearity limit of 9 μg/mL). An IgG titer equal or higher than 0.1 IU/mL for diphtheria and tetanus and higher than 10 mIU/mL for HBV (anti-HBs antibody titer) will be considered protective. An anti-HBs titer higher than 100 IU/mL will be considered to confer long-lasting protection
Correlation between quantification of relevant immune cells of HSCT recipients and vaccine response | at 3, 12 and 24 months after full block vaccination
  the association between blood T- B- and NK cell counts and subtypes of T and B cells (cells /mm3 of whole blood) and vaccine response will be analyzed
Correlation between proliferative T-cell response to mitogens and antigens and vaccine response | before and at 3 months after full block vaccination
  lymphocyte proliferation in response to ex vivo T cell stimulation (% of proliferating cells among CD3+ T-cells) will be evaluated The values measured will be defined as normal or abnormal, depending on whether they are within reference intervals (RI) derived from an independent set of healthy volunteers (REALISM protocol).
Correlation between innate immune response after ex vivo whole blood stimulation and vaccine response | before and at 3 months after full block vaccination
  The production of tumor necrosis factor (TNF) alpha released by blood cells in response to ex vivo stimulation by lipopolysaccharide (in pg/mL) will be measured The values measured will be defined as normal or abnormal, depending on whether they are within reference intervals (RI) derived from an independent set of healthy volunteers (REALISM protocol).
proportion of HSCT recipients with adverse event after each vaccination including local and general reactions | 21 days after each vaccination
  local and general reactions will be monitored for 30 min after each vaccination. Recipients will be given a diary card to record occurrence and severity of specific local reactions at the injection site and specific general reactions for 21 days after each vaccine injection.
ancillary study of cellular and humoral response to one dose of tetravalent inactivated influenza vaccine (IIV) | 4 weeks after influenza vaccination.
  Hemagglutination-inhibition assay (HAI) will be used to measure serum level concentrations of specific antibodies to the four influenza strains included in the vaccine.
  Immunization will be defined by seroprotective antibody titers ≥ 1:40 and/or seroconversion (4-fold rise in antibody titers).
  T-cell responses elicited by IIV will be measured ex vivo by interferon-Gamma ELISpot assay and expressed as number of spot-forming-cells.
  T-cell responses will be correlated to influenza antibody production, as measured by hemagglutination-inhibition assay (HAI).
  Influenza vaccine response in allo-HSCT recipients will be compared to that observed in Healthy Volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Florence ADER, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hôpital de la Croix Rousse, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conrad A, Boccard M, Valour F, Alcazer V, Tovar Sanchez AT, Chidiac C, Laurent F, Vanhems P, Salles G, Brengel-Pesce K, Meunier B, Trouillet-Assant S, Ader F; Lyon HEMINF Study Group. VaccHemInf project: protocol for a prospective cohort study of efficacy, safety and characterisation of immune functional response to vaccinations in haematopoietic stem cell transplant recipients. BMJ Open. 2019 Feb 15;9(2):e026093. doi: 10.1136/bmjopen-2018-026093. PMID 30772864